CLINICAL TRIAL: NCT03647397
Title: Use of PECO Air Purification in Hospital Rooms to Improve Health Outcomes for Pediatric Respiratory Distress
Brief Title: PECO Air Purification in Hospital Rooms to Improve Health Outcomes for Pediatric Respiratory Distress
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Molekule (Industry)
Collaborators: Mercy Health System (Network)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: Molekule-08082018
Record Dates: First submitted 2018-08-20; First posted 2018-08-27 (Actual); Last update posted 2019-05-17 (Actual); Status verified 2019-05

CONDITIONS: Asthma; Pneumonia; Respiratory Distress Syndrome
Keywords: asthma; environmental intervention; respiratory distress; pediatric hospitalization; pneumonia; bronchiolitis
MeSH Terms: conditions — Asthma; Pneumonia; Respiratory Distress Syndrome; Dyspnea; Bronchiolitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PECO (Experimental): All pediatric patients admitted for respiratory distress will have the intervention of Photo Electrochemical Oxidation (PECO) for Air Purification.
  Interventions: Device: Photo Electrochemical Oxidation (PECO) for Air Purification

INTERVENTIONS:
Device: Photo Electrochemical Oxidation (PECO) for Air Purification — PECO air purifiers from Molekule will be placed in every patient room. Health metrics will be tracked for patients whose diagnosis is respiratory distress.

SUMMARY:
This study will investigate the efficacy of a novel air purification technology, Photo Electrochemical Oxidation (PECO), has on pediatric patients hospitalized for respiratory distress. The study will take place at Mercyhealth Hospital - Rockton Avenue where all 23 pediatric rooms will be outfitted with portable PECO air purifying units. The main outcomes are the length of stay and progression to ICU, which will be compared with historical controls.

DETAILED DESCRIPTION:
The goal of this study is to assess whether using PECO to purify air in a hospital can improve health outcomes for pediatric patients with respiratory distress.

The results of this study will be used in three primary ways:

1. As evidence to support an installation of PECO in hospital HVAC systems to improve the standard of care for patients with respiratory distress
2. Towards dissemination efforts through publication in a peer-reviewed journal and presentation at national and international conferences
3. For informing healthcare providers and stakeholders

There are no plans to repeat this study with other hospital partners

ELIGIBILITY:
Inclusion Criteria: All pediatric patients who are admitted to the Mercyhealth Hospital - Rockton Avenue following the Start Date and have infectious or non-infectious respiratory distress as defined by the following ICD codes will be included in the study:

* J00-J06: Acute upper respiratory infections
* J09-J18: Influenza and pneumonia
* J20-J22: Other acute lower respiratory infections
* J30-J39: Other diseases of upper respiratory tract
* J40-J47: Chronic lower respiratory diseases
* J60-J70: Lung diseases due to external agents
* J80-J84: Other respiratory diseases principally affecting the interstitium
* J85-J86: Suppurative and necrotic conditions of the lower respiratory tract
* J90-J94: Other diseases of the pleura
* J95-J95: Intraoperative and postprocedural complications and disorders of respiratory system, not elsewhere classified

Exclusion Criteria:

* Any patient admitted to the NICU
* Patients in the ER only
* Any patient with non-respiratory conditions
* Adults

Ages: 1 Year to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 274 (Actual)
Dates: Start 2018-08-08 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Length of stay | 5 months
  Total length of hospital stay for patient

SECONDARY OUTCOMES:
Readmission rate | 1 months
  Rate of readmission within 30 days of discharge

CONTACTS AND LOCATIONS:
Overall Officials: Nikhil Rao, Principal Investigator — Molekule
Locations (1):
- Mercyhealth Hospital - Rockton Avenue, Rockford, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol (2018-10-10): https://cdn.clinicaltrials.gov/large-docs/97/NCT03647397/Prot_003.pdf